CLINICAL TRIAL: NCT07163689
Title: TIPS for the Management of Complicated Portal Hypertension Related to Porto-Sinusoidal Vascular Disease
Brief Title: TIPS for Complicated Portal Hypertension Related to Porto-Sinusoidal Vascular Disease
Acronym: TIPS-PSVD
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other); CHU Rennes (Unknown); AP-HP - HU BEAUJON (Unknown); University Hospital, Toulouse (Other); CHRU TOURS (Unknown); Centre Hospitalier Universitaire de Besancon (Other); Hospices Civils de Lyon, France (Unknown); APHP - HOPITAL AVICENNE (Unknown); University Hospital, Montpellier (Other); Saint-Luc University Hospital (Unknown); CHU Poitiers (Unknown); CHU NICE (Unknown); CH HENRI MONDOR (Unknown); Saint Antoine University Hospital (Other); University Hospital, Rouen (Other); AP-HP Paul Brousse University Hospital (Unknown); Nantes University Hospital (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Bordeaux (Other); University Hospital, Brest (Other); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0102
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: TIPS; Portal Hypertension; Porto-Sinusoidal Vascular Disease; Refractory Ascite; Esophageal Varices; Gastrointestinal Hemorrhage
Keywords: TIPS; Portal hypertension; Porto-Sinusoidal Vascular disease; refractory ascite; esophageal varices; gastrointestinal hemorrhage
MeSH Terms: conditions — Hypertension, Portal; Idiopathic Noncirrhotic Portal Hypertension; Esophageal and Gastric Varices; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group TIPS-PSVD: experimental group
- TIPS-cirrhose: historical control group

SUMMARY:
Porto-sinusoidal Vascular Disease (PSVD) is characterized by a portal hypertension (PH) without cirrhosis. This can induce PH complications, like digestive hemorrhage from esophageal or gastric varices, ascites, or even portal thrombosis. Due to the rarity of MVPS, the treatment of complications of portal hypertension is modeled on the methods used in cirrhotic portal hypertension with non-cardio-selective beta blockers, endoscopic ligations or diuretics in first line therapy, as proposed by the Baveno VII recommendations. In complicated or refractory forms of PH in PSVD, the place of TIPS is also discussed, as in the field of cirrhosis. However, the experience of TIPS in PSVD is limited, reported in case reports and small specifically dedicated series. No predictive factors for survival or recurrence and tolerance were well known. A larger study with control group is needed in order to better know the right time and the right indication for the use of TIPS in complicated PH PSVD-related.

The study will be retrospective, multicentric involving tertiary university French centers, expert in the management of TIPS. Patients white TIPS-PSVD will be compared with historical patients with TIPS-cirrhose, matched on age, sexe, indication of TIPS. The study will not comprise new intervention, only observational in a real life condition

ELIGIBILITY:
Inclusion Criteria:

* PSVD group :
* Patient with PSVD according VALDIG criteria
* TIPS for digestive hemorrhage on portal hypertension
* TIPS for refractory ascite
* TIPS for portal vein thrombosis
* Cirrhosis group with PH : (appaired by age, sexe, type of PH complications)
* Confirmed cirrhosis with :
* TIPS for digestive hemorrhage on portal hypertension
* TIPS for refractory ascite
* TIPS for portal vein thrombosis

Exclusion Criteria:

* no PSVD confirmed diagnosis
* Budd Chiari syndrome
* Rendu Osler disease; Heart failure
* Fontan; Sarcoïdosis
* Schistosomiase
* Congenitale liver fibrosis
* Abernathy syndrome
* Tumor infiltration by lymphoma
* Bone graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be retrospective and observational, collecting data provided in 24 tertiary french University Hospital (CHU).
  All patients with PSVD with a PH and treated by TIPS will be included (group TIPS_PSDV) and compared with an historical group of patients with Cirrhosis with a TIPS (group TIPS-cirrhose).
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
overall survival after TIPS placement | at 3 months
overall survival after TIPS placement | at 6 months
overall survival after TIPS placement | at 1 year
overall survival after TIPS placement | at 2 years
overall survival after TIPS placement | at 3 years
overall survival after TIPS placement | at 4 years
overall survival after TIPS placement | at 5 years

SECONDARY OUTCOMES:
free portal hypertension hemorrhage recurrence survival | at 3 months
free portal hypertension hemorrhage recurrence survival | at 6 months
free portal hypertension hemorrhage recurrence survival | at 1 year
free portal hypertension hemorrhage recurrence survival | at 2 years
free portal hypertension hemorrhage recurrence survival | at 3 years
free portal hypertension hemorrhage recurrence survival | at 4 years
free portal hypertension hemorrhage recurrence survival | at 5 years
free ascite recurrence survival | at 3 months
free ascite recurrence survival | at 6 months
free ascite recurrence survival | at 1 year
free ascite recurrence survival | at 2 years
free ascite recurrence survival | at 3 years
free ascite recurrence survival | at 4 years
free ascite recurrence survival | at 5 years
free TIPS dysfunction survival | at 3 months
free TIPS dysfunction survival | at 6 months
free TIPS dysfunction survival | at 1 year
free TIPS dysfunction survival | at 2 years
free TIPS dysfunction survival | at 3 years
free TIPS dysfunction survival | at 4 years
free TIPS dysfunction survival | at 5 years
complication of TIPS placement at D0 | at 3 months
complication of TIPS placement at D0 | at 6 months
complication of TIPS placement at D0 | at 1 year
complication of TIPS placement at D0 | at 2 years
complication of TIPS placement at D0 | at 3 years
complication of TIPS placement at D0 | at 4 years
complication of TIPS placement at D0 | at 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No